CLINICAL TRIAL: NCT00319072
Title: Testing an Interactive Website for Hormone Replacement
Brief Title: Hormone Replacement Therapy (HRT) Website Tool
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: AG0065; R44AG019082-03 (NIH)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2006-04

CONDITIONS: Communication; Menopause; Hormone Replacement Therapy
MeSH Terms: conditions — Communication

INTERVENTIONS:
Behavioral: TalkToYourDoc(sm) hormone therapy module

SUMMARY:
The purpose of this study is to evaluate a prototype web-based module for patients to generate appropriate and focused health information along with a customized set of questions to take to their health care provider for discussion on hormone replacement therapy.

DETAILED DESCRIPTION:
Patient-centered care may be enhanced by medically accurate, personalized health information generated by specialized software on the Internet. This study assessed the effect of a web-based interactive tool about menopausal hormone therapy (HT) on patient and provider communication and satisfaction.

The controlled, randomized evaluation of the TalkToYourDoc(sm) (TTYD) interactive website module on communication, satisfaction and efficiency of office visits involved 288 women born between 1930 and 1960 and 26 health care providers in an outpatient, academic setting. Women were randomized after stratification by HT use to usual care or access to the TTYD website. The TTYD website built a personalized series of questions based on participant input regarding health status and generated a printout of health issues, medications and questions about HT for participants to bring to the visit with their health care provider.

Results of the study found that women who participated in the intervention were more likely to come prepared to the clinic appointment with appropriate questions (80% vs. 96%) than women receiving usual care. Participants found the website easy to use, the questions generated were useful in the discussion of HT, and they felt that providers had a positive response to the printout. Providers felt that women who participated in the intervention were more engaged in the discussion and asked more relevant questions regarding HT. Providers had a higher level of satisfaction with the discussion with intervention participants, and felt that these office visits were more efficient.

Therefore, it was determined that the TalkToYourDoc(sm) module enhanced communication between women and their providers, led to greater visit satisfaction for both patient and provider, and improved visit efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Women born between 1930 to 1960
* Scheduled appointment at the OB/GYN or Family and Community Medicine out-patient clinics between 11/9/2004 to 12/2/2005

Exclusion Criteria:

* Men
* Current pregnancy
* Diagnosed cancer

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2004-03; Study Completion 2005-12

PRIMARY OUTCOMES:
Communication and satisfaction parameters from post-visit surveys of both patients and providers.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Eaker, ScD, Principal Investigator — Eaker Epidemiology Enterprises, LLC; Vanessa M. Barnabei, MD, PhD, Study Director — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Mechanic D. Physician discontent: challenges and opportunities. JAMA. 2003 Aug 20;290(7):941-6. doi: 10.1001/jama.290.7.941. PMID 12928472
- [Background] Mechanic D, McAlpine DD, Rosenthal M. Are patients' office visits with physicians getting shorter? N Engl J Med. 2001 Jan 18;344(3):198-204. doi: 10.1056/NEJM200101183440307. PMID 11172143
- [Background] Anderson GL, Limacher M, Assaf AR, Bassford T, Beresford SA, Black H, Bonds D, Brunner R, Brzyski R, Caan B, Chlebowski R, Curb D, Gass M, Hays J, Heiss G, Hendrix S, Howard BV, Hsia J, Hubbell A, Jackson R, Johnson KC, Judd H, Kotchen JM, Kuller L, LaCroix AZ, Lane D, Langer RD, Lasser N, Lewis CE, Manson J, Margolis K, Ockene J, O'Sullivan MJ, Phillips L, Prentice RL, Ritenbaugh C, Robbins J, Rossouw JE, Sarto G, Stefanick ML, Van Horn L, Wactawski-Wende J, Wallace R, Wassertheil-Smoller S; Women's Health Initiative Steering Committee. Effects of conjugated equine estrogen in postmenopausal women with hysterectomy: the Women's Health Initiative randomized controlled trial. JAMA. 2004 Apr 14;291(14):1701-12. doi: 10.1001/jama.291.14.1701. PMID 15082697
- [Background] Heisler M, Bouknight RR, Hayward RA, Smith DM, Kerr EA. The relative importance of physician communication, participatory decision making, and patient understanding in diabetes self-management. J Gen Intern Med. 2002 Apr;17(4):243-52. doi: 10.1046/j.1525-1497.2002.10905.x. PMID 11972720
- [Background] Martin LR, DiMatteo MR, Lepper HS. Facilitation of patient involvement in care: development and validation of a scale. Behav Med. 2001 Fall;27(3):111-20. doi: 10.1080/08964280109595777. PMID 11985184
- See also: The Benton Foundation — http://www.benton.org